CLINICAL TRIAL: NCT07111897
Title: Plate Fixation Versus Percutaneous Cannulated Screw Insertion in Sanders Type II and Type III Calcaneal Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS297/2025
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-05

CONDITIONS: Calcaneus Fractures
MeSH Terms: interventions — Fracture Fixation, Internal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percutaneous Cannulated Screws (Experimental)
  Interventions: Procedure: percutaneous cannulated screw fixation
- Plate Fixation (Experimental): Fixation of calcaneal fracture by plate
  Interventions: Procedure: Plate fixation

INTERVENTIONS:
Procedure: percutaneous cannulated screw fixation — fixation of calcaneal fractures by cannulated screws inserted percutaneously
  Arms: Percutaneous Cannulated Screws
Procedure: Plate fixation — Fixation of calcaneal fracture by plate.
  Other Names: osteosynthesis
  Arms: Plate Fixation

SUMMARY:
Sanders Ⅱ and Ⅲ intra-articular calcaneal fractures primarily result from falls from height, often accompanied by severe flap soft tissue injury and notable displacement of fracture fragments, which can pose significant reconstruction challenges. The traditional "L" lateral incision open reduction and internal fixation technique is considered the gold standard for the surgical treatment of calcaneal fractures. This trial aims to demonstrate that Percutaneous Cannulated Screws are not inferior to open reduction and internal fixation (ORIF) with plates in the treatment of calcaneal fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with calcaneal fractures according to Sanders classification are Sanders type II or type III.
2. Closed calcaneal fracture.
3. Patients aged 18-60.

Exclusion Criteria:

1. Patients with calcaneal fractures classified as Sanders type I or IV.
2. Open calcaneal fractures.
3. Patients with systemic comorbidities preventing surgical intervention (unfit patients).
4. Patients younger than 18 years old or older than 60.
5. Patients with associated spinal fractures.
6. Patients with other fractures in the same limb.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Bohler Angle | Preoperative, immediate postoperative, and at 6 months.
Gissane Angle | Preoperative, immediate postoperative, and at 6 months.
AOFAS Score | At 6 months.
Calcaneal width | Preoperative, immediate postoperative, and at 6 months.
Calcaneal height | Preoperative, immediate postoperative, and at 6 months.
Calcaneal length | Preoperative, immediate postoperative, and at 6 months.
Surgical time | intra-operative

SECONDARY OUTCOMES:
Time to union | at radiological evidence of healing, in 6 weeks.
Subtalar Arthritis | At 6 months.
Complication Rate | At 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Awab A. Moussa, MD Candidate, Study Director — Faculty of Medicine, Ain shams university, Cario, Egypt.
Locations (1):
- Faculty Of Medicine, Ain Shams university., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
For property rights and privacy protection

REFERENCES:
- [Background] 1. Rockwood Ca Jr, Greene DP. Rockwood and Green's fractures in adults. 4th ed. Philadelphia: Lippincott-Raven; 1996. p. 2405-62. 2. Mitchell MJ, McKinley JC, Robinson CM. The epidemiology of calcaneal fractures. Foot (Edinb). 2009 Dec;19(4):197-200. doi: 10.1016/j.foot.2009.05.001. PMID: 20307476. 3. Sanders R, Fortin P, DiPasquale T, Walling A. Operative treatment in 120 displaced intraarticular calcaneal fractures. Results using a prognostic computed tomography scan classification. Clin Orthop Relat Res. 1993 May;(290):87-95. PMID: 8472475IF: 4.2 Q1. 4. Yeo, J. H., Cho, H. J., & Lee, K. B. (2015). Comparison of two surgical approaches for displaced intra-articular calcaneal fractures: sinus tarsi versus extensile lateral approach. BMC musculoskeletal disorders, 16, 63. https://doi.org/10.1186/s12891-015-0519-0 5. Ibrahim T, Rowsell M, Rennie W, Brown AR, Taylor GJ, Gregg PJ: Displaced intra-articular calcaneal fractures: 15-year follow-up of a randomised controlled trial of conservative versus operative treatment. Injury 2007;38(7):848-855. 6. Gougoulias N, Khanna A, McBride DJ, Maffulli N: Management of calcaneal fractures: Systematic review of randomized trials. Br Med Bull 2009;92:153-167. 7. Swanson SA, Clare MP, Sanders RW: Management of intra-articular fractures of the calcaneus. Foot Ankle Clin 2008;13(4): 659-678. 8. Hsu AR, Anderson RB, Cohen BE. Advances in Surgical Management of Intra-articular Calcaneus Fractures. J Am Acad Orthop Surg. 2015 Jul;23(7):399-407. doi: 10.5435/JAAOS-D-14-00287IF: 2.6 Q1 . PMID: 26111874. 9. Backes, M., Schepers, T., Beerekamp, M. S., Luitse, J. S., Goslings, J. C., & Schep, N. W. (2014). Wound infections following open reduction and internal fixation of calcaneal fractures with an extended lateral approach. International orthopaedics, 38(4), 767-773. https://doi.org/10.1007/s00264-013-2181-1 10. Feng, Y., Shui, X., Wang, J. et al. Comparison of percutaneous cannulated screw fixation and calcium sulfate cement gra